CLINICAL TRIAL: NCT02373592
Title: Implementation of Foot Thermometry and SMS and Voice Messaging to Prevent Diabetic Foot Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: Johns Hopkins University (Other); Mayo Clinic (Other); University of Southern California (Other)
Responsible Party: Principal Investigator, Jaime Miranda, PhD, Universidad Peruana Cayetano Heredia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R21TW009982 (NIH)
Record Dates: First submitted 2015-02-20; First posted 2015-02-27 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-08

CONDITIONS: Diabetic Foot
Keywords: Diabetic Neuropathies; Thermometry; Diabetes Mellitus, Type 2; Foot Ulcer; Telemedicine
MeSH Terms: conditions — Diabetic Foot; Diabetic Neuropathies; Diabetes Mellitus, Type 2; Foot Ulcer | interventions — Spermine Synthase; Thermometry

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thermometry-only group (Placebo Comparator): Subjects will be provided with a TempStat (foot thermometer), a device that captures a thermal image of feet.
  Some alarm signs have been pre-specified: 1) thermal image shows yellow spots in any area of feet for two consecutive days, 2) thermal image shows different colors in contralateral areas of the feet for two consecutive days or, 3) a dermal lesion. In any of these three scenarios, subjects will be instructed to contact the study nurse by phone. (See Detailed Description for more detail on the actions after an alarm sign has been observed)
  Interventions: Device: Thermometry
- Thermometry plus SMS and voice messaging (Experimental): Thermometry-related intervention activities will be the same as those established for the thermometry-only group. In addition, this group will receive reminders to use the TempStat (two messages) and promote foot care (six messages). The content of these eight messages has been developed and validated through both SMS and voice messaging.
  During the first two weeks of the intervention, only reminders to use the TempStat will be sent, daily, Monday to Friday, both via SMS and voice messaging.
  Hereafter, for the remaining 76 weeks, patients will only receive two messages per week, one SMS and one voice message, alternating content (reminders to use TempStat and promotion of foot care).
  Interventions: Behavioral: SMS and voice messaging; Device: Thermometry

INTERVENTIONS:
Behavioral: SMS and voice messaging — This group will receive reminders to use the TempStat (two messages) and promote foot care (six messages). The content of these eight messages have been developed and validated their delivery through both, SMS and voice messaging.
  During the first two weeks of the intervention, only reminders to use the TempStat will be sent, daily, Monday to Friday, both via SMS and voice messaging.
  Hereafter, for the remaining 76 weeks, patients will only receive two messages per week, one SMS and one voice message, alternating content (reminders to use TempStat and promotion of foot care).
  Arms: Thermometry plus SMS and voice messaging
Device: Thermometry — Subjects will be provided with a TempStat (foot thermometer), a device that captures a thermal image of feet. (See Detailed description)

SUMMARY:
This study aims to implement daily temperature measurements of feet complemented by SMS and voice messaging to prevent diabetic foot ulcers in patients with type 2 diabetes mellitus at high risk of ulceration.

Design: Physician-blinded, randomized, 18-month trial.

Setting: Diabetes outpatient clinics from two public hospitals

Population: Subjects will be eligible if they (1) have a diagnosis of type 2 diabetes mellitus, (2) are between 18 - 80 years of age, (3) have a present dorsalis pedis pulse in both feet, (4) are in risk group 2 or 3 using the diabetic foot risk classification system as specified by the International Working Group on the Diabetic Foot, (5) have an operating cell phone or a caregiver with an operating cell phone, and (6) have the ability to provide informed consent.

Hypothesis: The investigators hypothesize that implementation of an enhanced intervention that combines daily temperature measurement for the reduction of diabetic foot ulcer with SMS and voice messaging will improve patient measurement compliance and reduce diabetic foot ulcers in a middle income country.

DETAILED DESCRIPTION:
Detailed Description:

Thermometry is a promising emerging modality for the prevention of diabetic foot ulcers according to different clinical trials. However, patient compliance with self-monitoring temperature at home is a concern, as they may be forgetful or find it difficult to get into a consistent routine of daily monitoring. Therefore, the investigators propose to determine the utility of SMS and voice messaging to remind the patients to perform the thermometry, and to assess the impact on diabetic foot ulceration.

Specific Aims are:

1. Compare the incidence of diabetic foot ulceration during the study between the arm that receives thermometry alone and the arm that receives thermometry plus SMS and voice messaging.
2. Compare the compliance with foot thermometer use between the two study arms.
3. Compare the frequency of alarms signs reported to the study nurse in the two study arms.
4. Compare the frequency of alarms signs reported in the patient's logbooks in the two study arms.
5. Compare the incidence of diabetic foot ulceration according to pre-specified sub-groups: caregiving status, and use of insoles and/or orthopedic shoes.
6. In the intervention-only group, compare the incidence of diabetic foot ulcers by varying the recipient of the messaging intervention (patient vs caregivers).

Intervention:

1. Placebo Comparator: Thermometry-only group. Subjects will be provided with a TempStat (foot thermometer), a device that captures a thermal image of feet through colors.

   Some alarm signs have been pre-specified: 1) When the thermal image shows yellow spots in any area of any feet for two consecutive days, 2) when the thermal image shows different colors in contralateral areas of the feet for two consecutive days or, 3) a dermal lesion is detected at any time. In any of these three scenarios, subjects will be instructed to contact the study nurse by phone or text message.

   For the first two types of alarm signs, once the study nurse is contacted he/ she will ask about the presence of lesions in the patient's feet and the patient's activity on the previous two weeks, and will provide recommendations on how to decrease activity until temperatures normalize. If TempStat measurements continue to show alarm signs for more than one week after the telephone consultation, the participant will be asked to contact the nurse and schedule a face-to-face evaluation to assess the presence of an infection and/or ulcer with a masked assessor.

   In the third type of alarm sign, presence of a dermal lesion, participants will be asked to contact the study's nurse and he/she will make an appointment for an evaluation with a nurse blind to the intervention.

   When the main outcome, foot ulceration, has been confirmed, patients will be directed by the study nurse to receive professional care by a specialist.
2. Experimental: Thermometry plus SMS and voice messaging Thermometry-related intervention activities will be the same as those established for the thermometry-only group. In addition, this group will receive reminders to use the TempStat (two messages) and promote foot care (six messages). The content of these eight messages has been developed and validated through both via SMS and voice messaging. During the first two weeks of the intervention, only reminders to use the TempStat will be sent, daily, Monday to Friday, both SMS and voice messaging. Hereafter, for the remaining 76 weeks, patients will only receive two messages per week, one SMS and one voice message, alternating content (reminders to use TempStat and promotion of foot care).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus.
* Dorsalis pedis pulse in both feet.
* In risk group 2 or 3 using the diabetic foot risk classification system as specified by the International Working Group on the Diabetic Foot.
* Operating cell phone or a caregiver with an operating cell phone.
* Ability to provide informed consent.

Exclusion Criteria:

* Current ulcers or open amputation sites.
* Active osteoarthropathy
* Severe peripheral vascular disease
* Foot infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Foot ulceration | 18 months
  The primary outcome is foot ulceration occurring at any point during the 12 month study duration.
  Foot ulceration will be defined using the American Diabetes Association criteria, which defines ulcers as any break in the cutaneous barrier; that usually extend through the full thickness of the dermis. There will be two ways of identifying if a patient has developed foot ulceration: (1) during the clinical evaluations done by a nurse every 2 months. (2) In addition to these bimonthly assessments, patients will be advised to make telephone calls to the study's nurse to report the presence of an ulcer, and he/she will be asked to go to the hospital for a face-to-face evaluation to be conducted by a masked nurse.

SECONDARY OUTCOMES:
Adherence to daily temperature measurement | 18 months
  Adherence to temperature measurements will be based on patient self-report of foot temperature monitoring through recording in patient's logbooks.
Report of an alarm sign to the nurse | 18 months
  Compare the frequency of alarms signs reported to the study nurse
Report of an alarm sign in the logbook | 18 months
  Compare the frequency of alarms signs reported in the patient's logbooks.
Dose-response analysis of SMS and voice messaging | 18 months
  Dose-response per protocol analysis will be performed.
Glycosilated hemoglobin control targets | 18 months
  Reduce of 1% or more of glycosylated hemoglobin.

OTHER OUTCOMES:
Sub-group analyses, all participants | 18 months
  The primary outcome will be subjected to pre-specified heterogeneity in treatment effects. In the following analyses, variables will be considered positive if its presence/usage is reported at baseline and in at the last evaluation of the participant during study period.
  1. Caregiving status, assistance provided to the patient with i) basic activities of daily living, or ii) in the identification, prevention, or treatment of diabetes or any disability.
  2. Use of insoles and/or orthopedic shoes.
Sub-group analyses, intervention group only | 18 months
  1)In order to receive the SMS and voice messaging, the intervention requires ownership of a cell phone by either the patient or its caregiver. This sub-group analysis will explore the primary outcome by the type of recipient (patient vs caregivers) of the messaging intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Miranda, MD, PhD, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (2):
- Peru (2):
  - Hospital Cayetano Heredia, Lima
  - Hospital Nacional Arzobispo Loayza, Lima

REFERENCES:
- [Background] Lazo-Porras M, Bernabe-Ortiz A, Sacksteder KA, Gilman RH, Malaga G, Armstrong DG, Miranda JJ. Implementation of foot thermometry plus mHealth to prevent diabetic foot ulcers: study protocol for a randomized controlled trial. Trials. 2016 Apr 19;17(1):206. doi: 10.1186/s13063-016-1333-1. PMID 27094007
- [Derived] Lazo-Porras M, Bernabe-Ortiz A, Taype-Rondan A, Gilman RH, Malaga G, Manrique H, Neyra L, Calderon J, Pinto M, Armstrong DG, Montori VM, Miranda JJ. Foot thermometry with mHeath-based supplementation to prevent diabetic foot ulcers: A randomized controlled trial. Wellcome Open Res. 2020 Aug 28;5:23. doi: 10.12688/wellcomeopenres.15531.2. eCollection 2020. PMID 32923686